CLINICAL TRIAL: NCT00374595
Title: Vascular Risk After Kidney Transplantation
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0053-95-FB; 1R01DK069919-01A2 (NIH)
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Results first posted 2023-08-09 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Cardiovascular Disease; Chronic Kidney Disease; Diabetes; Vitamin D Deficiency; Hyperparathyroidism
Keywords: Kidney Transplant; Vascular Risk; inflammation; Diabetes; Insulin resistance; Chronic kidney disease
MeSH Terms: conditions — Cardiovascular Diseases; Renal Insufficiency, Chronic; Diabetes Mellitus; Vitamin D Deficiency; Hyperparathyroidism; Inflammation; Insulin Resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypothesis: Nontraditional risk factors, such as inflammation, vitamin D deficiency, elevated PTH, insulin resistance, homocysteine, or uric acid, contribute to cardiovascular disease progression after kidney transplant.

The purpose of this study is to evaluate which traditional and nontraditional cardiovascular disease risk factors best predict progression of cardiovascular disease (CVD) using carotid intima media thickness performed by ultrasound, in kidney transplant patients.

DETAILED DESCRIPTION:
Cardiovascular disease remains the greatest cause of mortality after kidney transplant. Traditional risk factors, such as hypertension, diabetes, hyperlipidemia and smoking, contribute to vascular disease after transplant, but nontraditional risk factors may play a bigger role in vascular disease progression in this setting. This observational study will evaluate nontraditional risk factors for their contributions to vascular disease progression as determined by carotid intima media thickness and history of vascular disease events over time. The study requires annual checks of blood, urine, history, and carotid ultrasound for carotid intima media thickness

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant more than 6 months ago
* 19 years or older

Exclusion Criteria:

* Estimated GFR <30
* Previous small bowel, or lung transplant
* Pancreas transplant less than 6 months ago
* Cancer or any condition that would change weight dramatically in the near future such as malabsorption.
* Willing to return for testing annually for 3 years
* Women who are pregnant

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Transplant Clinic patients
Sampling Method: Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2012-07-26 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Larsen, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Kidney Transplant Recipients: This observational study evaluated nontraditional risk factors for their contributions to vascular disease progression as determined by carotid intima media thickness and history of vascular disease events over time. The study requires annual checks of blood, urine, history, and carotid ultrasound for carotid intima media thickness.
Period: Overall Study
Arm/Group | Kidney Transplant Recipients
Started | 338
Completed | 268
Not Completed | 70
Not completed — Death | 23
Not completed — Withdrawal by Subject | 39
Not completed — Lost to Follow-up | 3
Not completed — too much time commitment | 1
Not completed — transfer care to other clinical site | 1
Not completed — relocation | 3

BASELINE CHARACTERISTICS:
Arm/Group | Kidney Transplant Recipients
Number analyzed (Participants) | 338
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147
  Male | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 325
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 31
  White | 300
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Carotid Intima Media Thickness (CIMT)
Description: CIMT was defined by ultrasound. The mean and standard error of a 3 year change in CIMT was assessed (between baseline and three year follow up).
Time Frame: 3 years (baseline and three year follow up)
Population: 264 participants had 3 year follow-up for Carotid intima media thickness.
Measure: Mean (Standard Error); unit: millimeters (mm)
Arm/Group | Kidney Transplant Recipients
Number analyzed (Participants) | 264
millimeters (mm) | 0.044 (0.006)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Kidney Transplant Recipients
All-Cause Mortality (participants affected / at risk) | 23/338
Serious Adverse Events (participants affected / at risk) | 0/338
Other Adverse Events (participants affected / at risk) | 0/338

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes